CLINICAL TRIAL: NCT07058623
Title: A Randomized Controlled Trial of Nurse-Led Telehealth Versus In-Person Consultations in Detecting Complications and Improving Recovery After Total Knee Replacement
Brief Title: Nurse-Led Telehealth vs In-Person Follow-Up After Total Knee Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Wong King Sum, Associated Nurse Consultant (O&T), Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKR-TEL-2025-TKOH
Record Dates: First submitted 2025-06-10; First posted 2025-07-10 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Arthroplasty, Replacement, Knee; Osteoarthritis, Knee
Keywords: Total knee replacement; Knee arthroplasty; Postoperative care; Nurse-led telehealth; Telemedicine nursing consultation; Telehealth follow-up; Orthopedic nursing; Surgical complication detection; Recovery after knee surgery; Patient satisfaction; Outpatient follow-up care; Digital health interventions; HA Go mobile application; Remote patient monitoring
MeSH Terms: conditions — Osteoarthritis, Knee; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group design in which participants are randomly assigned to one of two groups: the nurse-led telehealth consultation group or the traditional in-person nursing consultation group. Both groups receive follow-up care after total knee replacement surgery, and their outcomes will be compared to evaluate the effectiveness of telehealth versus in-person consultations.
  Randomization is performed using block randomization with concealed allocation to ensure balance between groups and minimize selection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-Led Telehealth Consultation (Experimental): Participants receive postoperative nursing follow-up via virtual consultations using the HA Go mobile app, a secure, hospital-approved telehealth platform. Nurses monitor recovery, assess for complications, provide education, and manage minor issues remotely. Consultations are scheduled 2 weeks post-surgery, with additional sessions as clinically indicated, lasting approximately 20-30 minutes each. Support is provided to assist patients unfamiliar with the technology. This arm tests the effectiveness of remote nursing care compared to traditional in-person visits.
  Interventions: Procedure: Nurse-Led Telehealth Consultation
- Traditional In-Person Nursing Consultation (Active Comparator): Participants attend face-to-face postoperative nursing consultations at the Specialist Outpatient Department. Nurses perform physical assessments, monitor recovery progress, detect complications, provide education, and manage minor issues in-person. Follow-up visits are scheduled 2 weeks after surgery, with additional visits as needed. Consultations typically last 20-30 minutes. This arm represents standard care and serves as the active comparator to the telehealth intervention.
  Interventions: Procedure: Traditional In-Person Nursing Consultation

INTERVENTIONS:
Procedure: Nurse-Led Telehealth Consultation — Participants receive scheduled postoperative nursing consultations delivered remotely via the HA Go mobile application, a secure, hospital-approved telehealth platform. Consultations occur approximately two weeks after total knee replacement surgery, with additional sessions arranged as clinically needed within the first month post-surgery. Each telehealth session lasts about 20 to 30 minutes and includes assessment of recovery progress, monitoring for complications, patient education, and guidance on rehabilitation exercises. Patients receive technical support to facilitate effective use of the telehealth platform. This intervention leverages virtual care technology to provide convenient, accessible nursing follow-up without requiring in-person clinic visits.
  Other Names: Telehealth Nursing Consultation; Virtual Nurse Consultation; Remote Nursing Follow-Up; Telemedicine Nursing Care; HA Go App Nursing Consultation; Remote Postoperative Nursing
  Arms: Nurse-Led Telehealth Consultation
Procedure: Traditional In-Person Nursing Consultation — Participants receive scheduled postoperative nursing consultations in person at the Specialist Outpatient Department. Each consultation lasts approximately 20 to 30 minutes and includes physical assessment, monitoring for complications, patient education, and rehabilitation guidance. Follow-up visits are typically scheduled two weeks after total knee replacement surgery, with additional visits as clinically indicated. This intervention represents standard postoperative nursing care delivered face-to-face.
  Other Names: Face-to-Face Nursing Consultation; In-Clinic Nursing Follow-Up; Standard Nursing Consultation; Outpatient Nursing Visit; Postoperative In-Person Nursing Care
  Arms: Traditional In-Person Nursing Consultation

SUMMARY:
Brief Summary

The goal of this clinical trial is to learn if nurse-led telehealth consultations can help detect complications and support recovery after total knee replacement surgery. The study will compare telehealth nursing consultations to traditional in-person nursing visits.

The main questions it aims to answer are:

* Can nurse-led telehealth detect post-surgery complications as well as or better than in-person consultations?
* Does telehealth nursing support better or equivalent recovery outcomes and patient satisfaction compared to in-person care?

Participants will:

* Be adults who had their first total knee replacement surgery.
* Receive follow-up care either through telehealth consultations using the HA Go mobile app or through traditional face-to-face nurse visits in the outpatient clinic.
* Attend scheduled consultations and provide information about their recovery and any complications they experience.
* Complete surveys about their satisfaction with the care they receive.

This study will help determine if telehealth nursing consultations can provide safe, effective, and convenient follow-up care for patients after knee replacement surgery, potentially improving access and reducing travel burdens.

DETAILED DESCRIPTION:
Detailed Description This study is a randomized controlled trial designed to evaluate the clinical effectiveness and feasibility of nurse-led telehealth consultations compared to traditional in-person nursing consultations for post-operative care following total knee replacement (TKR) surgery.

Background and Rationale Total knee replacement is a common surgical intervention for end-stage knee osteoarthritis, offering significant pain relief and improved function. Post-operative follow-up is essential to monitor recovery, detect complications early, and support rehabilitation. However, traditional in-person consultations can pose logistical challenges for patients, including mobility limitations, travel burden, and time constraints. Telehealth has emerged as a promising alternative by enabling remote clinical assessments and patient monitoring, especially amplified by recent advances and adoption during the COVID-19 pandemic.

While telehealth models led by physicians have been studied extensively, there is a relative lack of evidence regarding nurse-led telehealth consultations in the orthopedic post-operative setting. Nurses play a crucial role in patient education, symptom monitoring, and care coordination, making nurse-led telehealth a potentially efficient and scalable solution. This study aims to fill this gap by rigorously evaluating whether nurse-led telehealth consultations can detect complications and support recovery as effectively as standard in-person visits.

Study Design

This is an open-label, parallel-group randomized controlled trial with two arms:

* Intervention arm: Nurse-led telehealth consultations delivered via a secure, hospital-approved mobile platform (the HA Go app).
* Control arm: Traditional in-person nursing consultations conducted at the Specialist Outpatient Department (SOPD).

Randomization will be performed using computer-generated block randomization with allocation concealment ensured through sealed opaque envelopes. Blinded outcome assessment and data analysis will be conducted to minimize bias.

Participants The trial will enroll adult patients (≥18 years old) who undergo first-time unilateral total knee replacement surgery at Tseung Kwan O Hospital. Eligible participants must be medically stable for discharge, have access to the necessary technology for telehealth, and provide informed consent. Patients with revision surgery, bilateral TKR, severe systemic disease (ASA Class III or above), or insufficient technological capacity will be excluded.

Interventions

Nurse-Led Telehealth:

Participants randomized to the telehealth arm will receive scheduled virtual consultations through the HA Go app. Consultations will include remote symptom assessment, wound evaluation via video, patient education on recovery and rehabilitation exercises, and management of minor complications. An executive assistant will provide technical support to patients unfamiliar with the app.

In-Person Nursing Consultation:

Participants assigned to the control group will attend face-to-face follow-up visits at the SOPD, receiving standard nursing care including physical examinations, education, and complication management.

Outcome Assessments The primary outcome is the rate of timely detection and management of post-operative complications within four weeks post-surgery. Secondary outcomes include functional recovery (assessed by validated scales such as KOOS), patient satisfaction, healthcare utilization (unplanned readmissions and emergency visits), and cost-effectiveness analyses encompassing travel and consultation time savings.

Data Collection and Management Data will be collected prospectively via electronic medical records, patient questionnaires, and telehealth system logs. Missing data will be managed using multiple imputation techniques under the assumption of missing at random. Security and confidentiality will be maintained according to Hospital Authority policies, with data encrypted and access restricted to authorized study personnel.

Significance By rigorously comparing nurse-led telehealth to traditional care, this study will generate high-quality evidence to inform post-operative management in TKR patients. Positive findings could support wider implementation of nurse-led telehealth services, improving accessibility, reducing patient burden, and optimizing healthcare resources. This model may be generalizable to other orthopedic and chronic disease care pathways.

Trial Registration and Ethics The study will be registered prior to recruitment, with ethical approval obtained from the Hospital Authority Central Institutional Review Board. Participants will provide informed consent, and the trial will adhere to CONSORT and Good Clinical Practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Undergoing their first total knee replacement surgery
* Within 4 weeks after surgery
* Medically stable for discharge and suitable for home-based follow-up care
* Have access to a smartphone and internet (for telehealth participants)
* Able to communicate effectively in Cantonese
* Provide informed consent to participate in the study

Exclusion Criteria:

* Undergoing bilateral or revision total knee replacement surgery
* Require immediate or intensive medical attention post-surgery (e.g., severe infection, hospitalization over 7 days)
* Have severe systemic disease (ASA physical status classification III or higher)
* Lack the technical ability or resources to participate in telehealth consultations
* Unable to communicate effectively in Cantonese
* Undergoing surgeries other than first-time total knee replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Postoperative Complications Detected Within Four Weeks Following Total Knee Replacement | Within 4 weeks (28 days) post-surgery
  This outcome measures the total number of participants in whom any postoperative complications are identified and managed during the follow-up period. Complications include both major events (e.g., deep vein thrombosis, surgical site infections) and minor issues (e.g., swelling, delayed wound healing, pain requiring intervention). The detection is based on clinical assessment during nurse-led telehealth or traditional in-person consultations.

SECONDARY OUTCOMES:
Change in Functional Recovery as Measured by the Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline (pre-surgery) and 3 months post-surgery
  This outcome measures participants' functional recovery and pain levels using the KOOS questionnaire, which ranges from 0 (extreme symptoms) to 100 (no symptoms). Higher scores indicate better recovery and function.
The Chinese version of the Mobile Health App Usability Questionnaire (I-C-MAUQ) (Telehealth group) | Within 4 weeks after surgery - immediately after the first telehealth follow-up consultation
  Patient-reported usability of the mobile-health platform will be assessed in participants randomised to the telehealth arm using the Chinese version of the Mobile Health App Usability Questionnaire (I-C-MAUQ). The 18 items are summed and rescaled to 0-100; higher scores denote better perceived usability and satisfaction with the nursing consultation.
Patient Satisfaction with Nursing Consultation | Within 4 weeks post-surgery, following the first consultation
  A standardized Hospital Authority patient satisfaction survey for both groups. Higher scores indicate greater satisfaction with the nursing consultation.
Unplanned Hospital Readmissions within 28 Days Post-Surgery | 28 days post-surgery
  This outcome records the number of participants who have unplanned hospital readmissions within 28 days after total knee replacement surgery.
Number of Visits to Accident and Emergency (A&E) Department within 3 Months Post-Surgery | 3 months post-surgery
  This outcome counts participant visits to the A&E department related to postoperative complications or concerns within 3 months after surgery.
Direct out-of-pocket travel cost (HK $) | Day of the first follow-up consultation (within 4 weeks after surgery)
  Total patient-paid transport expenditure, including fares, parking fees, and tolls, incurred for the index post-operative follow-up consultation. The amount is reported per participant in Hong Kong dollars.
Total travel time to clinic (minutes) | Day of the first follow-up consultation (within 4 weeks after surgery)
  Round-trip door-to-door travel duration self-reported by each participant for the index post-operative follow-up consultation. One value in minutes is recorded for every participant.
Nursing preparation time before follow-up consultation (minutes) | Day of the first follow-up consultation (within 4 weeks after surgery)
  Clock time a nurse spends on preparatory tasks for a single post-operative follow-up consultation. These tasks include initiating or joining the telehealth platform, verifying patient identity and coaching the patient on system login. Record one value per consultation, rounded to the nearest whole minute.
Nursing face-to-face consultation time (minutes) | Day of the first follow-up consultation (within 4 weeks after surgery)
  Elapsed clock time from the nurse's first direct interaction with the patient, either in person or on telehealth video, until completion of chart documentation and termination of the encounter. One value in whole minutes is recorded for each consultation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tseung Kwan O Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Demographics and Baseline Data: Including age, sex, and pre-operative ASA status.
  Primary Outcome: Data on the detection of post-operative complications within four weeks.
  Secondary Outcomes: Knee Injury and Osteoarthritis Outcome Score (KOOS) results , Mobile Health App Usability Questionnaire (I-C-MAUQ) scores , patient satisfaction surveys , healthcare utilization (unplanned readmissions, A&E visits) , and cost-effectiveness data (travel/consultation time).
  Adherence Data: Participant attendance and completion rates for scheduled consultations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start Date:
  Data will be available beginning 6 months after the publication of the primary manuscript.
  Justification: This is a standard academic practice that allows the primary research team a fair and exclusive period to analyze and publish their main findings before sharing the data.
  End Date:
  Data will be available for five years following the study's completion date (as defined in this registry).
Access Criteria: Access will be granted to qualified academic researchers for legitimate research purposes. Approved requesters will receive the de-identified IPD set, Study Protocol, Statistical Analysis Plan (SAP), and a blank Informed Consent Form (ICF).
  To request access, researchers must submit a formal proposal to the Principal Investigator. All requests require review by the study team and final approval from the Hospital Authority Central Institutional Review Board (HA Central IRB). An executed data-sharing agreement is mandatory before data transfer. Upon full approval, data will be shared via a secure, encrypted method.

REFERENCES:
- [Result] Zhao R, Cheng L, Zheng Q, Lv Y, Wang YM, Ni M, Ren P, Feng Z, Ji Q, Zhang G. A Smartphone Application-Based Remote Rehabilitation System for Post-Total Knee Arthroplasty Rehabilitation: A Randomized Controlled Trial. J Arthroplasty. 2024 Mar;39(3):575-581.e8. doi: 10.1016/j.arth.2023.08.019. Epub 2023 Aug 11. PMID 37572720
- [Result] Windsor EN, Sharma AK, Gkiatas I, Elbuluk AM, Sculco PK, Vigdorchik JM. An Overview of Telehealth in Total Joint Arthroplasty. HSS J. 2021 Feb;17(1):51-58. doi: 10.1177/1556331620972629. Epub 2021 Feb 21. PMID 33967642
- [Result] Visperas AT, Greene KA, Krebs VE, Klika AK, Piuzzi NS, Higuera-Rueda CA. A Web-Based Interactive Patient-Provider Software Platform Does Not Increase Patient Satisfaction or Decrease Hospital Resource Utilization in Total Knee and Hip Arthroplasty Patients in a Single Large Hospital System. J Arthroplasty. 2021 Jul;36(7):2290-2296.e1. doi: 10.1016/j.arth.2021.01.037. Epub 2021 Jan 21. PMID 33581971
- [Result] Shan Y, Ji M, Xie W, Li R, Qian X, Zhang X, Hao T. Chinese Version of the Mobile Health App Usability Questionnaire: Translation, Adaptation, and Validation Study. JMIR Form Res. 2022 Jul 6;6(7):e37933. doi: 10.2196/37933. PMID 35793132
- [Result] Pitaro NL, Barbera JP, Ranson WA, Zubizarreta N, Poeran J, Chen DD, Moucha CS, Hayden BL. Evaluating Resource Utilization for In-Person and Virtual Joint Classes in Total Joint Arthroplasty: An Analysis of Attendance Patterns at a Large Metropolitan Health System. J Arthroplasty. 2022 Sep;37(9):1708-1714. doi: 10.1016/j.arth.2022.03.079. Epub 2022 Apr 1. PMID 35378234
- [Result] McKeon JF, Alvarez PM, Vajapey AS, Sarac N, Spitzer AI, Vajapey SP. Expanding Role of Technology in Rehabilitation After Lower-Extremity Joint Replacement: A Systematic Review. JBJS Rev. 2021 Sep 13;9(9). doi: 10.2106/JBJS.RVW.21.00016. PMID 34516463
- [Result] Hofmann UK, Hildebrand F, Mederake M, Migliorini F. Telemedicine in orthopaedics and trauma surgery during the first year of COVID pandemic: a systematic review. BMC Musculoskelet Disord. 2023 Feb 7;24(1):101. doi: 10.1186/s12891-023-06194-3. PMID 36750962
- [Result] Fahey E, Elsheikh MFH, Davey MS, Rowan F, Cassidy JT, Cleary MS. Telemedicine in Orthopedic Surgery: A Systematic Review of Current Evidence. Telemed J E Health. 2022 May;28(5):613-635. doi: 10.1089/tmj.2021.0221. Epub 2021 Aug 10. PMID 34375150
- [Result] Fabres Martin C, Ventura Parellada C, Herrero Anton de Vez H, Ordonez Urgiles CE, Alonso-Rodriguez Piedra J, Mora Guix JM. Telemedicine approach for patient follow-up after total knee and reverse total shoulder arthroplasty: a pilot study. Int J Comput Assist Radiol Surg. 2023 Mar;18(3):595-602. doi: 10.1007/s11548-022-02784-z. Epub 2022 Nov 23. PMID 36422767
- [Result] El Ashmawy AH, Dowson K, El-Bakoury A, Hosny HAH, Yarlagadda R, Keenan J. Effectiveness, Patient Satisfaction, and Cost Reduction of Virtual Joint Replacement Clinic Follow-Up of Hip and Knee Arthroplasty. J Arthroplasty. 2021 Mar;36(3):816-822.e1. doi: 10.1016/j.arth.2020.08.019. Epub 2020 Aug 15. PMID 32893060
- [Result] Bovonratwet P, Song J, LaValva SM, Chen AZ, Ondeck NT, Blevins JL, Su EP. Telemedicine in Arthroplasty Patients: Which Factors Are Associated With High Satisfaction? Arthroplast Today. 2024 Jan 2;25:101285. doi: 10.1016/j.artd.2023.101285. eCollection 2024 Feb. PMID 38261888
- [Result] American Academy of Orthopaedic Surgeons. (2024). Total knee replacement. OrthoInfo. Retrieved January 8, 2025, from https://orthoinfo.aaos.org/en/treatment/total-knee-replacement